CLINICAL TRIAL: NCT03640442
Title: Modified Ramped Position for Intubation of Obese Females: a Randomized Controlled Study
Brief Title: Modified Ramped Position for Intubation of Obese Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-107-2018
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Obesity; Anesthesia
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ramped position group (Experimental): In this group, induction of anesthesia will be performed in the modified ramped position.
  Interventions: Other: Modified ramped position
- Ramped position group (Active Comparator): In this group, induction of anesthesia will be performed in the ordinary ramped position.
  Interventions: Other: Ramped position

INTERVENTIONS:
Other: Modified ramped position — This position will be achieved using a special pillow. Shoulders will be elevated and neck will be extended to bring the breasts away from the laryngoscopy. The patient will be positioned so that the tip of the last spinous process (C7) will be at the edge of the pillow. The neck will be extended to the most possible range.
  Arms: Modified ramped position group
Other: Ramped position — This position will be achieved by elevation of the shoulders and the head elevation till achieving alignment of sternal notch and external auditory meatus
  Arms: Ramped position group

SUMMARY:
The aim of this work is to investigate the feasibility of using the modified a ramped position for intubation of obese females in comparison to the traditional ramped position.

DETAILED DESCRIPTION:
Adequate conditions for endotracheal intubation require appropriate positioning of head and neck. The sniffing position had been described as the most appropriate head position for endotracheal intubation. Sniffing position is achieved through two main components: flexion of the neck by 35° (achieved by head elevation) and extension of the head by 15° 2 to have the sternum at the same level of external auditory meatus 34. Sniffing position has the advantage of alignment of the three axes: oral, pharyngeal, and laryngeal axes for reaching the optimal laryngeal visualization.

In obese patients, it is recommended to put the patient in the ramped position (back-up position with the tragus of the ear is at the level of the suprasternal notch) in addition to the sniffing head-and-neck position. Some commercially available pillows were introduced to facilitate laryngoscopy in obese patients such as: Troop elevation pillow and Rapid airway management positioner.

In addition to difficult laryngeal visualization, another problem commonly confronts anesthetists during intubation of obese females; that is impedance of laryngoscopy by large breasts. This problem commonly hinders the intubation process and might lead to serious hypoxia. Most of the positions described in literature were concerned with facilitating laryngeal visualization. No position to the best of our knowledge was applied to aid the introduction of the laryngoscope in the presence of large breasts.

The investigators hypothesized that using a special pillow to achieve a modified ramped position (by slight extension of the neck) at the beginning of the laryngoscopy would bring the breasts away from the laryngoscope. After successful introduction of the laryngoscope in the oral cavity, the head will be elevated using a head rest to achieve ordinary ramped position if laryngeal visualization was not adequate.

The aim of this work is to investigate the feasibility of using the aforementioned modified ramped position for intubation of obese females in comparison to the traditional ramped position.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* obese (with body mass index above 30 kg per squared meter)
* Scheduled for surgery under general anesthesia.

Exclusion Criteria:

* Patients with scars in the face or neck.
* Edentulous patients.
* Patients with airway masses.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Incidence of difficult laryngoscopy | 5 minutes after induction of general anesthesia
  defined as "failure to insert the laryngoscope in the oral cavity due to large breast with the need to reposition the patient to insert the laryngoscope"

SECONDARY OUTCOMES:
Time of laryngoscopy | 5 minutes after induction of general anesthesia
  Time measured in seconds from handling the laryngoscope till insertion of the whole blade length into the oral cavity
Time till complete visualization of the vocal cords | 5 minutes after induction of general anesthesia
  Defined as the time measured in seconds from handling the laryngoscope till visualization of the vocal cords.
Oxygen saturation | 5 minutes after induction of general anesthesia
  Oxygen saturation measured by pulse oximeter as percentage.
End-tidal carbon dioxide | 5 minutes after induction of general anesthesia
  End-tidal carbon dioxide measured in mmhg by capnography
Heart rate | 5 minutes after induction of general anesthesia
  Heart rate measured as number of heart beats per minute
incidence of difficult mask ventilation | 5 minutes
  The incidence of difficult mask ventilation defined as the need for high force or the need for additional assistant for maintenance of adequate ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hasanin, Professor, Principal Investigator — Assistant professor of anesthesia
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasanin A, Tarek H, Mostafa MMA, Arafa A, Safina AG, Elsherbiny MH, Hosny O, Gado AA, Almenesey T, Hamden GA, Mahmoud M, Amin S. Modified-ramped position: a new position for intubation of obese females: a randomized controlled pilot study. BMC Anesthesiol. 2020 Jun 17;20(1):151. doi: 10.1186/s12871-020-01070-2. PMID 32552691